CLINICAL TRIAL: NCT00141713
Title: The Use of Etanercept (Enbrel®) in the Treatment of Acute Graft-Versus-Host Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Principal Investigator, John Levine, MD, Professor of Pediatrics, University of Michigan Rogel Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 3-37; 2003-0591 (Other: University of Michigan IRBMED); FD-R-002397-03-2 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2005-08-30; First posted 2005-09-01 (Estimated); Last update posted 2013-03-13 (Estimated); Status verified 2013-03

CONDITIONS: Graft-Versus-Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Etanercept

ARMS (1):
- 1 (Experimental): etanercept treatment for GVHD
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Etanercept — Patients enrolled on the study will receive etanercept at 0.4 mg/kg per dose up to a maximum of 25 mg per dose subcutaneously twice a week. Etanercept must be initiated within 72 hours of starting solumedrol.

SUMMARY:
Etanercept (Enbrel) will be added to standard therapy for acute Graft-versus-Host Disease to see if the effectiveness of standard therapy can be improved.

Partial Funding Source- FDA OOPD

DETAILED DESCRIPTION:
The standard treatment for acute graft-versus-host disease is a combination of steroids and tacrolimus or cyclosporine. Previous work has shown that less than 50% of patients respond fully to GVHD. Without a good response, patients often have a prolonged treatment for this disease, often involving hospitalization and sometimes even death.

Etanercept is a drug that blocks a chemical called Tumor Necrosis Factor (TNF) from causing damage to tissue. Etanercept (Enbrel) will be added to help improve the response to standard treatment for graft-versus-host disease (GVHD).

This is an experimental research project. It is not known whether the etanercept will actually improve the body's response to graft-versus-host disease. This treatment is meant to determine if etanercept will improve your response to treatment of GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patient may be transplanted with stem cells from any source using either a myeloablative or nonmyeloablative preparative regimen
* Patient may be any age
* Patient must have biopsy proven new onset of aGVHD; Clinical Grading must be II-IV and may occur after stem cell transplant or donor leukocyte infusion (DLI). Patients may begin Etanercept treatment prior to biopsy confirmation of GVHD. Acute GVHD will be determined by clinical presentation and not timing from stem cell infusion
* Patient must be on solumedrol at a dose of 2mg/kg/day of actual body weight for no more than 72 hours prior to the initiation of etanercept
* Patient must have evidence of neutrophil engraftment with an ANC of > 500 for three consecutive days
* Pulse ox > 90% on room air

Exclusion Criteria:

* Pregnancy or nursing mother
* Intolerance or allergic reaction to etanercept
* Previous use of steroids for treatment of acute GVHD
* Active infection, chronic or localized, not responding to antibiotics, with continued signs of infection (patients with a positive C. Difficile test will not be excluded from the study)
* Condition that might predispose to developing serious infections (i.e. active and uncontrolled diabetes mellitus, sickle cell anemia)
* Other investigational agents for the treatment or prophylaxis of graft-vs-host disease within the past 2 weeks
* Serum creatinine > 2.0mg/dl
* Patients being treated for acute pulmonary dysfunction (IPS) study using etanercept
* Patients with hypotension believed to be secondary to sepsis syndrome or heart failure requiring > 1 inotropic agent, or dopamine >5mcg/kg/minute for blood pressure support
* Evidence of congestive heart failure on clinical exam
* Evidence of hepatic dysfunction with an ALT or AST > 2.5 x ULN, not due to GVHD

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2003-10; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the response rate of etanercept when administered with steroids for treatment of biopsy proven aGVHD. | at 1, 2, and 3 months

SECONDARY OUTCOMES:
To analyze intracellular cytokine levels, lymphocyte phenotype and plasma cytokine levels in patients with aGVHD before and after treatment with etanercept and to correlate these laboratory endpoints with clinical outcomes during the trial. | at 1, 2, and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MS MD, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Levine JE, Paczesny S, Mineishi S, Braun T, Choi SW, Hutchinson RJ, Jones D, Khaled Y, Kitko CL, Bickley D, Krijanovski O, Reddy P, Yanik G, Ferrara JL. Etanercept plus methylprednisolone as initial therapy for acute graft-versus-host disease. Blood. 2008 Feb 15;111(4):2470-5. doi: 10.1182/blood-2007-09-112987. Epub 2007 Nov 27. PMID 18042798